CLINICAL TRIAL: NCT06949761
Title: A Phase Ib/II Clinical Study to Evaluate the Safety, Tolerability, and Efficacy of QLC1101 in Combination With Other Therapies in the Treatment of Patients With Advanced Solid Tumors Harboring a KRAS G12D Mutation
Brief Title: A Clinical Study to Evaluate the Safety, Tolerability, and Efficacy of QLC1101 in Combination With Other Therapies in the Treatment of Patients With Advanced Solid Tumors Harboring a KRAS G12D Mutation
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QLC1101-201
Record Dates: First submitted 2025-04-22; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- QLC1101+QL1203 (Experimental)
  Interventions: Drug: QLC1101+QL1203
- QLC1101+QL2107 (Experimental)
  Interventions: Drug: QLC1101+QL2107
- QLC1101+QL1706 (Experimental)
  Interventions: Drug: QLC1101+QL1706
- QLC1101+docetaxel (Experimental)
  Interventions: Drug: QLC1101+docetaxel

INTERVENTIONS:
Drug: QLC1101+QL1203 — QLC1101 is an innovative small molecule inhibitor targeting KRAS G12D with independent intellectual property rights developed by Qilu Pharmaceutical Co., Ltd.；QL1203, developed by Qilu Pharmaceutical Co., Ltd., is a recombinant anti-EGFR fully human monoclonal antibody injection and a biosimilar to Vectibix®
  Arms: QLC1101+QL1203
Drug: QLC1101+QL2107 — QLC1101 is an innovative small molecule inhibitor targeting KRAS G12D with independent intellectual property rights developed by Qilu Pharmaceutical Co., Ltd.；QL2107 developed by Qilu Pharmaceutical Co., Ltd. is a potential biosimilar to Pembrolizumab (Keytruda®)
  Arms: QLC1101+QL2107
Drug: QLC1101+QL1706 — QLC1101 is an innovative small molecule inhibitor targeting KRAS G12D with independent intellectual property rights developed by Qilu Pharmaceutical Co., Ltd.；QL1706 Injection (QL1706) is a combination antibody developed by Qilu Pharmaceutical Co., Ltd. It consists of two full-length immunoglobulin G (IgG) antibodies: anti-PD-1 monoclonal antibody (hereafter referred to as anti-PD-1) and anti-CTLA-4 monoclonal antibody (hereafter referred to as anti-CTLA-4)
  Arms: QLC1101+QL1706
Drug: QLC1101+docetaxel — QLC1101 is an innovative small molecule inhibitor targeting KRAS G12D with independent intellectual property rights developed by Qilu Pharmaceutical Co., Ltd.；Docetaxel is a tubulin binding agent that prevents cell division by stabilizing microtubule structure and leads to apoptosis
  Arms: QLC1101+docetaxel

SUMMARY:
A Phase Ib/II Clinical Study to Evaluate the Safety, Tolerability, and Efficacy of QLC1101 in Combination with Other Therapies in the Treatment of Patients With Advanced Solid Tumors Harboring a KRAS G12D Mutation.

The study includes Phase Ib (combination therapy with dose escalation stage) and Phase II (expansion stage). The study will includes a total of 4 cohorts:

Phase Ib will enroll subjects in 4 cohorts (cohorts 1-4). Subjects will be allocated to appropriate cohorts by the investigator according to specific indications and treated with the corresponding combination regimen for safety and tolerability assessment. The Bayesian optimal interval (BOIN) design will be used for dose escalation and MTD determination.

In Phase II, according to the results of the Phase Ib and SMC decision, 1-2 appropriate dose groups will be selected. In the dose group(s), the sample size (including subjects in the dose escalation stage) will be increased to 20 for each indication according to the cohort for expansion to further evaluate the efficacy of QLC1101 combination therapy in the treatment of subjects with advanced solid tumors harboring KRAS G12D mutations

ELIGIBILITY:
Inclusion Criteria:

* Subjects confirmed advanced (metastatic or unresectable) solid tumors with KRAS G12D mutations.
* Subjects who have failed or are unable to tolerate standard therapy, have no standard therapy, or refuse to receive standard therapy
* The investigator confirms that the subject has at least one measurable lesion recorded by CT and/or MRI according to RECIST v1.1
* ECOG PS score: 0 or 1

Exclusion Criteria:

* Subjects who have been previously treated with inhibitors for KRAS G12D mutations
* Subjects with known immediate or delayed hypersensitivity or idiosyncratic reaction to the components of the drug products used in the study
* Subjects with known or symptomatic active central nervous system (CNS) metastases or carcinomatous meningitis at screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
adverse events | from first dose to 90 days after last dose
  any untoward medical occurrence in a subject who received an investigational product, which can be manifested as any symptoms, signs, diseases, or laboratory test abnormalities, and do not necessarily have a causal relationship with the investigational product